CLINICAL TRIAL: NCT06354361
Title: A Randomized Control Trial Examining the Efficacy of a Novel, Trauma-informed Approach to Cognitive Remediation (Goal Management Training) in Public Safety Personnel With Post-traumatic Stress Disorder (PTSD) and Co-morbid Conditions
Brief Title: Trauma-Informed Goal Management Training for Public Safety Personnel (PSP) With Post-traumatic Stress Disorder (PTSD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Workplace Safety and Insurance Board (Unknown)
Responsible Party: Principal Investigator, Margaret McKinnon, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17440
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Goal Management Training (GMT); Trauma-Informed Goal Management Training (TI-GMT)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into two groups.
  One group will receive nine sessions of Trauma-Informed Goal Management Training, and the other group will receive nine sessions of standard Goal Management Training.
  Each group session will be 2 hours long, and offered virtually (using Zoom for Healthcare).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma-Informed GMT (TI-GMT; offered online) (Experimental): Participants randomly assigned to the TI-GMT condition will be asked to attend nine weekly, 2-hour virtual group sessions of TI-GMT via Zoom for Healthcare, a PHIPA-compliant video conferencing platform. Each group will consist of 1 or 2 facilitators and up to 10 participants.
  Interventions: Behavioral: Trauma-Informed Goal Management Training (TI-GMT)
- Standard GMT (GMT; offered online) (Active Comparator): Participants randomly assigned to the GMT condition will be asked to attend nine weekly, 2-hour virtual group sessions of GMT via Zoom for Healthcare, a PHIPA-compliant video conferencing platform. Each group will consist of 1 or 2 facilitators and up to 10 participants.
  Interventions: Behavioral: Goal Management Training (GMT)

INTERVENTIONS:
Behavioral: Trauma-Informed Goal Management Training (TI-GMT) — Trauma Informed-Goal Management Training (TI-GMT) is a modified version of Goal Management Training (GMT), a cognitive remediation program that emphasises mindfulness and practice in planning and completing goal-oriented behaviours. TI-GMT enhances the standard GMT protocol with the addition of several trauma-informed adaptations and content that is sensitive and specific to public safety personnel with PTSD.
  Participants are trained to interrupt ongoing disruptive behaviours through the resumption of executive control to help define goal hierarchies and monitor goal achievement. Mindfulness meditation helps develop attentional control and the skill of bringing one's mind to the present. Real-life examples are incorporated to illustrate goal attainment failures and successes, and participants practice solving complex, real-life tasks in sessions.
  Sessions include instructional material, interactive tasks, discussion of real-life deficits, and homework/practice activities.
  Arms: Trauma-Informed GMT (TI-GMT; offered online)
Behavioral: Goal Management Training (GMT) — Goal Management Training (GMT) is a cognitive remediation program that emphasises mindfulness and practice in planning and completing goal-oriented behaviours.
  Participants are trained to interrupt ongoing disruptive behaviours through the resumption of executive control to help define goal hierarchies and monitor goal achievement. Mindfulness meditation helps develop attentional control and the skill of bringing one's mind to the present. Real-life examples are incorporated to illustrate goal attainment failures and successes, and participants practice solving complex, real-life tasks in sessions.
  Sessions include instructional material, interactive tasks, discussion of real-life deficits, and homework/practice activities.
  Arms: Standard GMT (GMT; offered online)

SUMMARY:
Goal Management Training (GMT) is a program designed to help improve cognitive functioning. For this study, researchers have worked closely with the developers of this program to create a modified version called Trauma-Informed Goal Management Training (TI-GMT), that is more sensitive to the needs of public safety personnel (PSP) diagnosed with Post-Traumatic Stress Disorder (PTSD).

The goal of this clinical trial is to find out how effective this modified, Trauma-Informed Goal Management Training program is for public safety personnel diagnosed with Post-Traumatic Stress Disorder, in comparison to the standard Goal Management Training program.

The main questions it aims to answer are:

1. Does Trauma-Informed Goal Management Training result in better neuropsychological functioning and greater reductions in the severity of PTSD symptoms when compared to standard Goal Management Training?
2. Does Trauma-Informed Goal Management Training result in self-reported improvements in cognitive functioning and the overall ability to function (including intent to return to work, and/or intent to stay at work, reductions in disability status, etc.) when compared to standard Goal Management Training?
3. Does Trauma-Informed Goal Management Training continue to benefit individuals three months after treatment?

Participants will:

* complete three separate assessments before starting the treatment - a clinical interview to evaluate symptoms, a cognitive assessment, and completing a set of questionnaires
* participate in a nine-week group treatment program (one day a week for two hours)
* complete three separate assessments after completing the treatment - a clinical interview to evaluate symptoms, a cognitive assessment, and completing a set of questionnaires
* complete three separate assessments three months after completing the treatment - a clinical interview to evaluate symptoms, a cognitive assessment, and completing a set of questionnaires

ELIGIBILITY:
Inclusion Criteria - participants must:

* be fluent in English
* reside in Ontario
* be public safety personnel (e.g. police officer, corrections officer, probation or parole officer, firefighter, search and rescue, paramedic, nurse, dispatcher)
* be able to provide written informed consent
* meet criteria on the PTSD Checklist for DSM-5 (PCL-5) for a provisional diagnosis of PTSD (cut-off score of >30), administered during screening
* be able to attend regular online, 2-hour sessions once a week for 9 weeks, and be willing to complete the pre- and post- treatment assessments
* have access to a smart phone, tablet, or computer with a working microphone and camera, and have reliable and consistent internet

Exclusion Criteria:

* daily or almost daily use of benzodiazepines
* daily or almost daily use of narcotics
* diagnosed with alcohol use disorder OR substance use disorder in the past 12 months
* meet criteria on the Mini-International Neuropsychiatric Interview (M.I.N.I.) for diagnosis of alcohol use disorder OR substance use disorder
* history of moderate-to-severe brain injury and/or loss of consciousness with prolonged effects that interfere with daily functioning at school, work, or family unit
* history of neurological disorder(s) that may impact ability to participate in the study
* diagnosis of psychotic disorder(s) or bipolar disorder(s)
* diagnosis of neurodevelopmental disorder(s) that may impact ability to participate in the study
* other conditions/impairments/considerations that may interfere with completion of study tasks
* previous participation in Goal Management Training
* receiving treatment with anti-cholinergic medication, anti-psychotic medication, or psychostimulants
* had electroconvulsive therapy (ECT) within the past year
* currently engaged in a trauma-specific intervention that may impact the findings of the current study such as Eye Movement Desensitization and Reprocessing (EMDR), Cognitive Processing Therapy (CPT), Prolonged Exposure (PE), etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symptom severity as assessed by the Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders-5th Edition ('CAPS-5') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 30-item structured, clinician-administered interview used to make a lifetime or current diagnosis of PTSD and to assess PTSD symptoms.
  Questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms on social and occupational functioning, and specifications for the dissociative subtype.
  Total scores for severity may range between 0 and 80, with higher scores indicating greater symptom severity.
Change from baseline in scores on the Sustained Attention Response Task ('SART') subtest of the Creyos Battery at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 'game-ified' Go/No-Go task that assesses sustained attention, this task requires participants to inhibit a behavioural response to a single, infrequent target appearing amidst a presentation of frequent non-targets.
  This task will be administering remotely, using Zoom for Healthcare (a PHIPA-compliant video conferencing platform) and Creyos (a web-based platform for assessing cognitive functioning).
  Scores are calculated based on accuracy of responses (errors) and reaction time (reaction time variability and slowing after errors). Higher scores on each indicate more errors, more variability in reaction time, and more slowing after an error, respectively.
  A percentile rank ranging between 1 and 99 is generated to indicate the individual's performance in comparison to a population of individuals of the same gender and age group.

SECONDARY OUTCOMES:
Demographic Information | Collected at baseline only
  Age, sex, race, education, relationship status, employment status, and profession (whether police, firefighter, volunteer firefighter, search and rescue personnel, paramedic, nurse, correctional officer, probation officer, parole officer, or emergency dispatcher).
Scores on the Life Events Checklist for Diagnostic and Statistical Manual of Mental Disorders-5th Edition ('LEC-5') at baseline | Administered at baseline only
  A self-report measure designed to screen for potentially traumatic events in a respondent's lifetime by assessing exposure to 16 events known to potentially result in PTSD or distress, as well as one additional item to assess any other extraordinarily stressful event not captured in the first 16 items.
  There is no formal scoring protocol or interpretation, as this measure simply identifies whether a person has experienced one or more of the events listed.
Scores on the Childhood Trauma Questionnaire ('CTQ') at baseline | Administered at baseline only
  A self-report measure that assesses for exposure to five forms of common childhood trauma -- sexual abuse, physical abuse, emotional abuse, physical neglect, emotional neglect.
  All sub-scales (or, the five forms of childhood trauma) have a possible score range of 5 to 25.
  Higher scores reflect greater exposure to childhood trauma.
Scores on the Advanced Clinical Solutions ('ACS') Test of Premorbid Functioning ('TOPF') at baseline | Administered at baseline only
  The Advanced Clinical Solutions (ACS) Test of Premorbid Functioning (TOPF) provides an estimate of pre-morbid intellectual functioning, and will be administered using Zoom for Healthcare (a PHIPA-compliant video conferencing platform).
  The test yields one raw score (total number of words correctly read before the discontinue criteria was met) that is converted to a T score. Higher T scores indicate better performance on this task.
Change from baseline in scores on the Mini International Neuropsychiatric Interview 7.0.2 ('M.I.N.I.') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A structured clinician-administered interview that assesses psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition. Diagnostic modules utilised:
  i) Major Depressive Episode ii) Suicidality iii) Manic and Hypomanic Episodes iv) Panic Disorder v) Agoraphobia vi) Social Anxiety Disorder vii) Obsessive Compulsive Disorder viii) Alcohol Use Disorder ix) Substance Use Disorder x) Psychotic Disorders and Mood Disorder with Psychotic Features xi) Anorexia Nervosa xii) Bulimia Nervosa; xiii) Binge Eating Disorder xiv) Generalized Anxiety Disorder
  This is a diagnostic clinical interview; scores are not reported on a scale.
Change from baseline in scores on selected neuropsychological assessment measures of Executive functioning, Processing speed and Attention at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  The Double Trouble, Feature Match, Spatial Planning, and Odd One Out subtests of the 'Creyos' battery will be administered remotely using Zoom for Healthcare (a PHIPA-compliant video conferencing platform) and 'Creyos' (a web-based platform for assessing cognitive functioning) to assess executive functioning, processing speed, and attention.
  A standard score (mean=100, SD=15) and corresponding percentile rank are derived from the individual's raw score to indicate where the individual's scores fall on a normal distribution. An individual with a standard score of 100 and corresponding percentile rank of 50 is exactly at the average score for these tasks, and scores above or below 100 can easily be understood in relation to this average. Higher scores may indicate greater performance on these tasks.
  Hypothetically, under the normal distribution, the 'minimum' and the 'maximum' values are unbounded, however, in practice, these values may range between ≤ 20 and ≥ 150.
Change from baseline in scores on the California Verbal Learning Test (CVLT-3) at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  The California Verbal Learning Test (CVLT-3, standard and alternate forms) will be administered over PHIPA-compliant video conferencing as an assessment of declarative memory.
  Scaled scores (mean=10, SD=3), ranging between 1 and 19, and corresponding percentile ranks, are derived from the individual's raw scores to indicate where the individual's scores fall on a normal distribution.
  Higher scores on correctly recalled items indicate greater performance on these tasks; higher scores in recall errors may reflect greater deficits.
Change from baseline in scores on selected neuropsychological assessment measures of Declarative memory at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  Declarative memory will also be assessed using the Paired Associates and Digit Span subtests of the 'Creyos' battery (a web-based platform for assessing cognitive functioning) over PHIPA-compliant video conferencing.
  A standard score (mean=100, SD=15) and corresponding percentile rank are derived from the individual's raw score to indicate where the individual's scores fall on a normal distribution. An individual with a standard score of 100 and corresponding percentile rank of 50 is exactly at the average score for these tasks, and scores above or below 100 can easily be understood in relation to this average. Higher scores on correctly recalled items indicate greater performance on these tasks; higher scores in recall errors may reflect greater deficits.
  Hypothetically, under the normal distribution, the 'minimum' and the 'maximum' values are unbounded, however, in practice, these values may range between ≤ 20 and ≥ 150.
Change from baseline in scores on selected neuropsychological assessment measures of Intellectual functioning at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  The Grammatical Reasoning subtest of the 'Creyos' Battery will be administered remotely using PHIPA-compliant video conferencing and 'Creyos' (a web-based platform for assessing cognitive functioning) as an assessment of the ability to quickly understand and make valid conclusions about concepts expressed in words.
  A standard score (mean=100, SD=15) and corresponding percentile rank are derived from the individual's raw score to indicate where the individual's scores fall on a normal distribution. An individual with a standard score of 100 and corresponding percentile rank of 50 is exactly at the average score for these tasks, and scores above or below 100 can easily be understood in relation to this average. Higher scores may indicate greater performance on these tasks.
  Hypothetically, under the normal distribution, the 'minimum' and the 'maximum' values are unbounded, however, in practice, these values may range between ≤ 20 and ≥ 150.
Change from baseline in scores on selected neuropsychological assessment measures of Visuospatial and Visuoconstructive Ability and Sensorimotor integration at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  The Rotations (mental manipulation of visual stimuli) and Polygons (visuospatial processing) subtests of the 'Creyos' Battery will be administered remotely using PHIPA-compliant video conferencing and 'Creyos' (a web-based platform for assessing cognitive functioning) to assess visuospatial and visuoconstructive ability and sensorimotor integration.
  A standard score (mean=100, SD=15) and corresponding percentile rank are derived from the individual's raw score to indicate where the individual's scores fall on a normal distribution. An individual with a standard score of 100 and corresponding percentile rank of 50 is exactly at the average score for these tasks, and scores above or below 100 can easily be understood in relation to this average. Higher scores may indicate greater performance on these tasks.
  Hypothetically, under the normal distribution, the 'minimum' and the 'maximum' values are unbounded, however, in practice, these values may range between ≤ 20 and ≥ 150.
Change from baseline in scores on selected neuropsychological assessment measures of Visual and Visuospatial Working Memory at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  Token Search (visual working memory), Monkey Ladder (visuospatial working memory), and Spatial Span (spatial short-term memory) subtests of the 'Creyos' Battery will be administered remotely using PHIPA-compliant video conferencing and 'Creyos' (a web-based platform for assessing cognitive functioning) to assess visual and visuospatial working memory.
  A standard score (mean=100, SD=15) and corresponding percentile rank are derived from the individual's raw score to indicate where the individual's scores fall on a normal distribution. An individual with a standard score of 100 and corresponding percentile rank of 50 is exactly at the average score for these tasks, and scores above or below 100 can easily be understood in relation to this average. Higher scores may indicate greater performance on these tasks.
  Hypothetically, under the normal distribution, the 'minimum' and the 'maximum' values are unbounded, however, in practice, these values may range between ≤ 20 and ≥ 150.
Change from baseline in score on the Depression and Anxiety Stress Scale ('DASS-21') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A self-report measure that assesses the presence and severity of symptoms of depression, anxiety, and stress over the last week.
  Respondents rate their symptoms on a 4-point scale with 0 representing absence of the symptom and 3 representing a symptom occurring almost all the time. Three scores are computed, one for each sub-scale (depression, anxiety, and stress), by summing all the values of the items on each respective sub-scale.
  Higher scores reflect greater symptom severity; calculated scores can be used to qualify the severity of the symptoms (e.g., normal/minimal, mild, moderate, severe, extremely severe).
Change from baseline in score on the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5th Edition ('PCL-5') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 20-item self-report measure that assesses the severity of PTSD symptoms according to the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders-5th Edition.
  Symptom domains are intrusions, avoidance, negative alterations in mood and cognitions, and alterations in arousal and reactivity.
  A total score, ranging between 0 and 80, is derived by summing all the values of the items, and a cut-off point of 33 is suggested to indicate a probable PTSD diagnosis.
Change from baseline in score on the Multiscale Dissociation Inventory ('MDI') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 30-item self-report measure that assesses six domains of dissociative symptoms over the past month -- disengagement, depersonalisation, derealisation, emotional constriction, memory disturbance, and identity dissociation.
  A total score, ranging between 30 and 150, is derived by summing all the values of the items; higher total scores indicate greater dissociation.
Change from baseline in score on the Difficulties in Emotion Regulation Scale ('DERS') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 36-item self-report measure that assesses difficulties with emotion regulation across six domains -- nonacceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.
  Higher scores may indicate greater dysfunction in emotion regulation.
Change from baseline in score on the twenty-item Toronto Alexithymia Scale ('TAS-20') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 20-item self-report measure that assesses difficulties recognising and naming emotions across three domains -- difficulty identifying feelings, difficulty describing feelings, and externally oriented thinking.
  Individuals with scores less than or equal to 51 are interpreted as having no alexithymia, individuals with scores between 52 and 60 are interpreted as having possible alexithymia, and individuals with scores greater than or equal to 61 are interpreted as having alexithymia.
Change from baseline in score on the Moral Injury Assessment for Public Safety Personnel ('MIA-PSP') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 17-item self-report measure of work-related morally injurious experiences unique to public safety personnel across three underlying factors -- perpetrations, betrayals, and emotional sequelae.
  Higher scores reflect greater exposure to morally injurious experiences.
Change from baseline in scores on the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 75-item standardised self-report measure that captures an individual's views of their executive functions or self-regulation in their everyday environment across nine non-overlapping theoretically and empirically derived clinical scales:
  Inhibit, Self-Monitor, Plan/Organise, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organisation of Materials.
  Responses to items are summed up to generate raw scores, which are then converted to T scores. Higher T scores typically reflect greater difficulties in the corresponding aspects of executive dysfunction.
Change from baseline in scores on the Cognitive Failures Questionnaire 2.0 ('CFQ 2.0') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 15-item self-report measure that captures subjective experiences of cognitive failures in daily life. Each item is rated on a Likert scale from 0 ("Never") to 4 ("Very often").
  Higher scores may indicate greater self-reported impairment in cognitive functioning.
Change from baseline in scores on the Return to work Obstacles and Coping Efficacy - Common Mental Disorders ('ROSES-CMD') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  Evaluates obstacles participants may face when returning to work (part A) and how capable they feel they are of overcoming them (part B).
  Items use a 7-point response scale and include specific questions to assess perceived obstacles and self-efficacy beliefs about overcoming the obstacles.
  Higher scores on 'obstacles' items and lower scores on 'self-efficacy' items indicate decreased readiness to return-to-work.
Change from baseline in scores on the World Health Organization's Disability Assessment Schedule ('WHODAS 2.0') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A 36-item self-report measure that assesses health and disability on six domains of functioning:
  cognition, mobility, self-care, getting along (interacting with others), life activities, and participation (participating in society).
  Higher values may indicate greater functional impairment.
Change from baseline in scores on the Lam Employment Absence and Productivity Scale ('LEAPS') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  A self-report measure designed to assess and monitor work functioning and productivity.
  Participants are asked to respond to 4 questions; the fourth question assesses specific symptoms by having participants respond to 7 sub-questions on a 5-point scale.
  Two values of interest for this study are derived:
  i) measure of work impairment (sum of responses to the 7 sub-questions) ii) percent of work hours missed due to impairment [raw score of item 3 (hours of work missed) divided by raw score of item 2 (hours of work scheduled) multiplied by 100].
  A total score, ranging from 0-28, is derived by summing responses to the 7 sub-questions; higher scores indicate greater work impairment.
Change from baseline in scores on the Survey of Perceived Organizational Support ('SPOS') at post-intervention and follow-up | Baseline, post-intervention at 9 weeks, and 3-month follow-up
  An 8-item survey that assesses the extent to which an individual believes that their organisation is
  1. committed to them,
  2. values their continued membership, and
  3. is generally concerned about their well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McKinnon, PhD, Principal Investigator — McMaster University

REFERENCES:
- [Background] Boyd JE, O'Connor C, Protopopescu A, Jetly R, Rhind SG, Lanius RA, McKinnon MC. An Open-Label Feasibility Trial Examining the Effectiveness of a Cognitive Training Program, Goal Management Training, in Individuals With Posttraumatic Stress Disorder. Chronic Stress (Thousand Oaks). 2019 Apr 18;3:2470547019841599. doi: 10.1177/2470547019841599. eCollection 2019 Jan-Dec. PMID 32440592
- [Background] Protopopescu A, O'Connor C, Cameron D, Boyd JE, Lanius RA, McKinnon MC. A Pilot Randomized Controlled Trial of Goal Management Training in Canadian Military Members, Veterans, and Public Safety Personnel Experiencing Post-Traumatic Stress Symptoms. Brain Sci. 2022 Mar 12;12(3):377. doi: 10.3390/brainsci12030377. PMID 35326333
- [Background] Boyd JE, Sanger BD, Cameron DH, Protopopescu A, McCabe RE, O'Connor C, Lanius RA, McKinnon MC. A Pilot Study Assessing the Effects of Goal Management Training on Cognitive Functions among Individuals with Major Depressive Disorder and the Effect of Post-Traumatic Symptoms on Response to Intervention. Brain Sci. 2022 Jun 30;12(7):864. doi: 10.3390/brainsci12070864. PMID 35884671